CLINICAL TRIAL: NCT01001182
Title: Rheumatoid Arthritis in Greece: The Economic Burden of the Disease and the Impact on Quality of Life
Brief Title: Health Outcomes in Rheumatoid Arthritis in Greece
Acronym: HORA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A1-102329; B1801120
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
Keywords: observational; non-interventional; prospective
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non interventional: Patients with RA diagnosis receiving any treatment for RA (DMARDS or biologics)
  Interventions: Other: non interventional

INTERVENTIONS:
Other: non interventional — non interventional

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic debilitating disease, causing severe pain and progressive joint destruction and leading to partial loss of mobility. The disease has a severe impact on patients' quality of life, due to the pain and physical impairment it causes, which can also result in psychological and social difficulties. Moreover, the chronic nature of the disease deems necessary the long-term use of medication, causing significant costs to the patient and the healthcare system. The decline in functional ability can cause problems at work, with reduced productivity or even unemployment. In addition, RA can limit the patients' ability for self-care, hence imposing a further burden on the patients' families and the society.

Many international studies have confirmed the reduced quality of life for people suffering from RA [1-3], as well as the large economic impact of the disease on the patients, the health system and society [4-6]. However, no assessment of the above impact of RA on the Greek population has been published so far.

A wide research of the literature confirms the relationship between costs and quality of life on the one hand and functional ability (as measured by the Health Assessment Questionnaire) on the other hand. [7-8] The impact of functional ability on quality of life is straightforward, however studies also demonstrate that as disease symptoms progress, without proper treatment, the overall costs undertaken by the patient or the healthcare system can rise significantly. On the other hand, if effective treatment can lessen or postpone the most serious consequences of the disease (such as extensive joint damage that could lead to surgical replacement), the savings on healthcare can offset some of the costs of the more effective drug therapies.

In the light of the above findings, it seems important that in order to properly assess therapeutic strategies for RA patients it is necessary to have an accurate view of the total burden of RA on the population. It is also important to be able to establish a robust relationship between functional ability and impact of RA on costs and quality of life.

DETAILED DESCRIPTION:
The study will use a prevalence-based approach, recruiting patients at various stages of disease. Subjects will be enrolled sequentially as per their order of appearance at the site, until the maximum allowed number of subjects is reached at each site.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older
* Confirmed diagnosis of theumatoid arthritis by investigating physician.
* Evidence of a personally signed and dated informed consent document (or legally acceptable representative).

Exclusion Criteria:

* Simultaneous participation in an interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older with confirmed RA diagnosis will be included in the study. The investigating physician must confirm RA diagnosis during the patient's visit.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Quality of life | 1 year
Resource utilization | 1 year
Productivity losses | 1 year

SECONDARY OUTCOMES:
Functional ability | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Greece (7):
  - Pfizer Investigational Site, Alexandroupoli, Alexandroupoli
  - Pfizer Investigational Site, Athens, Athens
  - Pfizer Investigational Site, Heraklion, Crete
  - Pfizer Investigational Site, Ioannina, Ioannina
  - Pfizer Investigational Site, Mezourlo, Larissa
  - Pfizer Investigational Site, Rio, Patras
  - Pfizer Investigational Site, Thessaloniki, Thessaloniki

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-102329&StudyName=Health%20Outcomes%20in%20Rheumatoid%20Arthritis%20in%20Greece